CLINICAL TRIAL: NCT06416722
Title: Multidimensional Evaluation of the Effectiveness of Telerehabilitation-Based Dual-Task Training in Parkinson's Patients
Brief Title: Telerehabilitation Dual-Task Training for Parkinson's: A Multidimensional Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Ezgi Gul, MSc, PT, Research Asistant, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 28.03.2024/ 59
Record Dates: First submitted 2024-05-11; First posted 2024-05-16 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cognitive-Motor Dual Task Activities Group (Experimental): Patients included in this group will be given additional cognitive tasks.
  Interventions: Other: Cognitive-Motor Dual Task Activities
- Motor-Motor Dual Task Activities Group (Experimental): Patients included in this group will be given additional motor tasks.
  Interventions: Other: Motor-Motor Dual Task Activities
- Cognitive-Motor & Motor-Motor Dual Task Activities Group (Experimental): Simultaneously with balance and large amplitude functional activities.
  Interventions: Other: Cognitive-Motor & Motor-Motor Dual Task Activities

INTERVENTIONS:
Other: Cognitive-Motor Dual Task Activities — Patients included in this group will be given additional cognitive tasks (e.g. counting months, subtracting 5 from 100) in accordance with the physiotherapist's commands simultaneously with balance and large amplitude functional activities (such as stepping forward-sideways-backwards, sitting and standing).
  Arms: Cognitive-Motor Dual Task Activities Group
Other: Motor-Motor Dual Task Activities — Patients included in this group will be given additional motor tasks (e.g. passing the ball from the right hand to the left hand while standing on a soft surface, clapping) in accordance with the physiotherapist's commands simultaneously with balance and large amplitude functional activities (such as stepping forward-sideways-backwards, sitting and standing).
  Arms: Motor-Motor Dual Task Activities Group
Other: Cognitive-Motor & Motor-Motor Dual Task Activities — Simultaneously with balance and large amplitude functional activities (such as stepping forwards-sideways-backwards, sitting and standing), patients included in this group will be given additional cognitive (e.g. counting while standing with feet closed) and motor (e.g. passing the ball from the right hand to the left hand while standing on a soft surface) tasks in accordance with the physiotherapist's commands.
  Arms: Cognitive-Motor & Motor-Motor Dual Task Activities Group

SUMMARY:
In this clinical study, the aim is to assess the effectiveness of telerehabilitation-based dual-task training in improving balance and gait function among individuals diagnosed with Parkinson's Disease. Parkinson's Disease is characterized by motor symptoms such as tremors and slowness of movement, as well as cognitive impairments. While medical treatments help manage symptoms, exercise programs are vital for enhancing physical and cognitive functions.

Dual-task training involves combining motor and cognitive activities to enhance gait and balance control, and recent studies have shown its effectiveness in Parkinson's Disease rehabilitation. However, there's limited research on delivering dual-task training through telerehabilitation and determining the optimal content for maximum benefits.

This project involves 30 Parkinson's Disease patients who will be randomly assigned to three groups receiving different dual-task exercise programs via telerehabilitation. Each program focuses on combining balance and functional exercises with either cognitive or motor secondary activities. The exercises will be performed three times a week for four weeks under the guidance of a physiotherapist via Zoom.

Before and after the intervention, participants will be evaluated for feasibility, gait, balance, cognition, and activity levels. Researchers of this study hypothesize that telerehabilitation-based dual-task training will significantly improve balance and gait function in Parkinson's Disease patients, offering a convenient and effective treatment option to enhance their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with idiopathic Parkinson's Disease
* Stage 1-3 on the Hoehn-Yahr scale
* A minimum score of 21 on the Montreal Cognitive Assessment Scale test
* Stable drug treatment within the last 1 month
* Patients are in the "On" period
* Ability to walk independently on level ground (3 and above according to Functional Ambulation Classification)

Exclusion Criteria:

* Serious hearing or vision problems
* Having other neurological, cardiovascular or orthopaedic disorders that may prevent walking
* Any other neurological disorder (e.g. dementia, cerebrovascular disease)
* less than 5 years of education
* To have vascular lower extremity pathologies
* Not having internet access via smartphone or computer

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility Assessment | Baseline and after the interventions (4th week)
  The study's feasibility will be assessed through various measures. Firstly, we'll assess Participation Rate by calculating the ratio of attended sessions to the total. Participants will provide reasons for missed sessions, and their feedback will be recorded. After each session, participants will rate their fatigue on the Borg Perceived Exertion Scale, aiming to keep effort levels moderate (scores 12-17). To evaluate difficulty, participants will rate dual-task exercises on a Visual Analog Scale (0-10). Higher scores indicate greater difficulty, averaged over the study. Finally, at the end of the four-week program, participant satisfaction will be evaluated using a telerehabilitation-based exercise program questionnaire.
Digit Span Test | Baseline and after the interventions (4th week)
  The Digit Span Test, consisting of forward and backward sequences, is administered separately. Each sequence comprises numbers with digits incrementing sequentially. Numbers are read aloud to the subject at a rate of one per second. Success in any trial prompts the initiation of the next trial. However, failure in both trials results in discontinuation of the test. The length of the last successfully repeated sequence determines the span range.
Mental Flexibility | Baseline and after the interventions (4th week)
  In the Mini-Mental State Examination, as part of the Attention and Calculation subsection, individuals are asked to subtract 7 repeatedly from 100, continuing until reaching 65. Those with five years of education or less who cannot complete this task are then asked to perform an alternative task: counting the days of the week starting from Sunday and counting backwards. In both assessments, one point is awarded for each correct operation.
Word Fluency Test | Baseline and after the interventions (4th week)
  This test is based on saying as many words that are not proper nouns or verbs beginning with the letters F, A, S as possible in one minute. One minute is given for each letter. The total score is equal to the total number of words uttered in all letters. It measures verbal-phonemic fluency. In the standardisation study conducted in our country, the letters K, A, S were used. In this study, the total number of words will be evaluated.
Gait Assessment | Baseline and after the interventions (4th week)
  Kinovea® version 0.8.15 software will be utilized to obtain objective and quantitative data for spatiotemporal parameters of gait (stride length, double stride length, support surface, stride width, cadence, walking speed, step duration) and kinematic parameters of gait. In the study, a 3-meter walking distance of the subjects will be recorded with a camera placed in the sagittal plane. Coloured marks will be placed on the right and left heels, and these marks will be tracked and annotated on the video. The obtained videos will be observed, and the parameters of stride length (the distance between two consecutive heel strikes of one limb and the other limb) and double stride length (the distance between two consecutive heel strikes of the same limb) will be analyzed independently with Kinovea motion analysis software.
Mini-BEST Test | Baseline and after the interventions (4th week)
  The Mini-BEST test, which will be used for dynamic balance assessment, is a 14-item balance scale and evaluates postural reactions, sensory orientation and dynamic walking sub-parameters. In the last part, it allows the assessment of dual-task performance within the scope of the Forced-Reach-Walk Test (with Cognitive Loading). Each item in the test is scored between (0-2); a score of 0 indicates that the person is unable to perform the task, while a score of 2 is normal. The total score will be between 0 and 28. The total score reflects the balance ability. Higher scores mean better balance ability. It is a valid and reliable measurement method that requires approximately 15 minutes to complete, is one-dimensional and valid for use in Parkinson's Disease.
Four-step square test | Baseline and after the interventions (4th week)
  The four-step square test is a clinical assessment used to evaluate the ability to change direction while stepping, particularly focusing on dynamic balance and mobility. During the test, the patient starts in the upper left square (Square 1) and faces Square 2. The step sequence initially moves clockwise: Square 1, then Squares 2, 4, and 3. Subsequently, the sequence reverses, moving anti-clockwise: Square 3, followed by Squares 4, 2, and back to Square 1. The physiotherapist demonstrates the test, allowing the patient to practice and learn the sequence. If the patient cannot complete the sequence successfully, loses balance, or touches a support cane, the test is repeated. Two scores are obtained, and the better of the two scores is recorded. Timing begins when the patient's first foot touches the floor in Square 2 and ends when their second foot touches the floor in Square 1. The shorter the time, the better the result for this test.
Postural Stability Assessment | Baseline and after the interventions (4th week)
  KFORCE Plates are a type of force platform utilized to objectively measure postural control parameters. These plates enable the assessment of both static and dynamic balance across a broad spectrum of movements. Consisting of two independent plates, they have the capability to determine weight distribution during the stance phase and calculate the center of gravity. KFORCE Plates evaluate various positions such as standing, single-leg stance, and squatting, providing a comprehensive report with multiple data points post-assessment. This assessment will significantly enhance the project by offering objective data on changes in postural control following exercise interventions and allowing for a more detailed interpretation compared to scale-based assessments.
Parkinson's Activity Scale | Baseline and after the interventions (4th week)
  Parkinson's Activity Scale, a scale developed to evaluate functional activities in Parkinson's Disease, provides information about the transfer status of patients. Scored between 0 and 4 points, a high score indicates good performance. The scale has subdivisions including getting up from a chair, in-bed mobilisation and gait akinesia. In this study, it will be used to evaluate the functional activity status of the patients. High score indicates good functional performance.
Dual Task Questionnaire | Baseline and after the interventions (4th week)
  The Dual Task Questionnaire consists of 10 questions designed to assess the frequency of difficulties associated with daily tasks involving dual tasking. It is used to measure how often individuals have problems with the content of the questionnaire. In response to the questions, individuals are asked to choose from five options ranging from very often to never or not applicable (5-point scale, using a 0-4 scale). The resulting score is divided by 10 for an average rating per question.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakırköy Prof. Dr. Mazhar Osman Ruh Sağlığı ve Sinir Hastalıkları Eğitim ve Araştırma Hastanesi, Istanbul, Bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No